CLINICAL TRIAL: NCT02922075
Title: Soft and Hard Tissue Stability After Immediate Tooth Replacement With Implant in Fresh Sockets Grafted With Different Soft Tissue Grafts
Brief Title: Impact of Soft Tissue Grafts on Tissue Alterations After Immediate Tooth Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: São Paulo State University (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: São Paulo State University
Record Dates: First submitted 2016-09-24; First posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Tooth Socket; Dental Implants
Keywords: gingival recession; immediate implant and provisional placement; bone graft; connective tissue graft; collagen matrix
MeSH Terms: conditions — Gingival Recession | interventions — Immediate Dental Implant Loading; Tooth Extraction; Bone Regeneration; Bio-Gide; Amoxicillin; Acetaminophen; Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CTL (Placebo Comparator): No soft tissue graft was used. It was performed tooth extraction, immediate implant, immediate restoration, bone regeneration, post operative medication and definitive prosthesis.
  Interventions: Device: Immediate implant; Procedure: Tooth extraction; Device: Immediate restoration; Biological: Bone regeneration; Drug: Post operative medication; Device: Definitive prosthesis; Other: No soft tissue graft
- CM (Experimental): Patient received a collagen matrix graft. It was performed tooth extraction, immediate implant, immediate restoration, bone regeneration, post operative medication and definitive prosthesis.
  Interventions: Biological: Collagen matrix graft; Device: Immediate implant; Procedure: Tooth extraction; Device: Immediate restoration; Biological: Bone regeneration; Drug: Post operative medication; Device: Definitive prosthesis
- CTG (Experimental): Patient received a connective tissue graft. It was performed tooth extraction, immediate implant, immediate restoration, bone regeneration, post operative medication and definitive prosthesis.
  Interventions: Biological: Connective tissue graft; Device: Immediate implant; Procedure: Tooth extraction; Device: Immediate restoration; Biological: Bone regeneration; Drug: Post operative medication; Device: Definitive prosthesis

INTERVENTIONS:
Biological: Connective tissue graft — A 1.5 mm thick soft tissue graft removed from the palate with determined dimensions. The recipient site was prepared by performing laterally a delicate elevation of the facial tissue avoiding the mesial and distal papilla. The soft tissue graft length was equal to the horizontal distance between the two papillas and its length was set at 6 mm. Soft tissue grafts were placed at the level of the gingival margin and stabilized with simple interrupted sutures.
  Other Names: autogenous subepithelial connective tissue graft
  Arms: CTG
Biological: Collagen matrix graft — A 15x20 mm collagen matrix trimmed according to determined dimensions. The recipient site was prepared by performing laterally a delicate elevation of the facial tissue avoiding the mesial and distal papilla. The soft tissue graft length was equal to the horizontal distance between the two papillas and its length was set at 6 mm. Soft tissue grafts were placed at the level of the gingival margin and stabilized with simple interrupted sutures.
  Other Names: heterogenous graft
  Arms: CM
Device: Immediate implant — A conical implant with a morse-taper connection with moderate roughness implant surface was properly installed in the ideal tridimensional position with its platform placed 4 mm below the facial gingival margin. After tooth extraction and dental implant installation with a torque > 32 Ncm patients were randomized into three groups (8 patients per group): 1- No soft tissue graft, Control group (CTL); 2- Collagen Matrix group (CM); 3- Connective tissue graft group (CTG).
Procedure: Tooth extraction — Compromised tooth was gently removed and the socket was debrided thoroughly, cleansed and inspected. The socket's palatal and apical bone was sequentially drilled. All surgeries were performed by the same surgeon and were individually planned according to the clinical and tomographic evaluation. Implant diameter was set as 3.5 mm and its length was selected according to the quantity of bone available apically to the fresh alveolar socket.
Device: Immediate restoration — A titanium abutment was installed in the dental implant with manual torque and a prefabricated tooth shell was relined with resin material to fabricate cement or screw retained interim restoration. All interim restorations were installed in infra-occlusion matching the adjacent teeth color and form, with light proximal contacts and presented a subgingival concave contour.
Biological: Bone regeneration — All sites received a non-cross linked collagen membrane and deproteinized bovine bone mineral containing 10% of porcine collagen.
  Other Names: Bio-Oss Collagen®; Bio-Gide®
Drug: Post operative medication — Postoperative instructions were given, antibiotics were prescribed for 7 days (amoxicillin 500 mg t.i.d), analgesics to relieve from pain (Paracetamol 750 mg) and chlorhexidine 0.12% rinse twice a day for 15 days. Complementary, the patients were instructed to avoid chewing in the anterior region and to follow a soft diet.
  Other Names: Amoxicillin; Paracetamol; Chlorhexidine
Device: Definitive prosthesis — Definitive implant-supported restorations were performed 6 months after dental implant placement.
  Other Names: Zirconia abutment and ceramic crown installation
Other: No soft tissue graft — No soft tissue graft was used
  Arms: CTL

SUMMARY:
This study evaluates the impact of soft tissue grafts on soft tissue recession following immediate implant, provisional and bone graft placement in compromised sockets. One third of the patients received a collagen matrix (CM group), another third received a connective tissue graft removed from the palate (CTG group) and the final third did not receive any soft tissue graft (CTL group).

DETAILED DESCRIPTION:
Preventing soft tissue recession following flapless immediate implant and provisional placement (IIPP) in sockets with facial bone dehiscences is a challenge, mainly in esthetic areas. This study evaluated the impact of soft tissue grafts on peri-implant alterations after 1-year follow-up. Twenty-four patients with one single failing maxillary incisor presenting facial bone dehiscence and receiving IIPP were randomly divided in three groups (n= 8 in each group): Control (CTL); Collagen Matrix (CM); Connective tissue graft (CTG). In addition to soft tissue grafts, all groups were treated with collagen membrane and deproteinized bovine bone mineral containing 10% of porcine collagen. Clinical, photographic and tomographic analyses were performed at baseline, 6 and 12 months after surgery to evaluate tissue alterations.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a failing maxillary incisor with neighbouring teeth and harmonic gingival contour;
* Operated area with appropriate palatal/apical bone to install the implant;
* A buccal wall defect confirmed by cone beam computed tomography;
* Clinical attachment level > 3 mm;
* Good oral hygiene with visible plaque index < 20%;
* No bone loss in the neighbouring teeth;
* Implant primary stability > 32N

Exclusion Criteria:

* History of periodontal surgeries in the failing tooth;
* Occlusal instability;
* Systemic alterations that could compromise the surgical procedure, such ass smokers, bruxists; drug users; patients with diabetes or pregnants.
* Active infection involving the gingival margin
* Patients undergoing radiotherapy in the head and neck area. Patients presented history of bone associated diseases or medication affecting bone metabolism;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Periimplant marginal recession | 12 months after surgical procedure
  Periimplant marginal recession in millimeters 12 months after the surgical procedure.

SECONDARY OUTCOMES:
Questionnaire of Implant survival | 12 months
  Evaluation of implant survival
Papilla migration | 12 months after the surgical procedure
  Evaluation of mesial and distal papilla migration in millimeters 12 months after the surgical procedure
Pink esthetic score | 12 months after the surgical procedure
  Evaluation of pink esthetic scores
Soft tissue thickness | 12 months after the surgical procedure
  Evaluation of soft tissue thickness in millimeters 12 months after the surgical procedure
Bone height | 12 months after the surgical procedure
  Evaluation of bone height in millimeters in contact with the implant 12 months after the surgical procedure
Modified pink esthetic score | 12 months after the surgical procedure
  Evaluation of gingival esthetics
Bone thickness | 12 months after the surgical procedure
  Evaluation of bone thickness in millimeters in contact with the implant 12 months after the surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Elcio Marcantonio Jr, Professor, Principal Investigator — Professor
Locations (1):
- Araraquara Dental School at the São Paulo State University, Araraquara, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yoshino S, Kan JY, Rungcharassaeng K, Roe P, Lozada JL. Effects of connective tissue grafting on the facial gingival level following single immediate implant placement and provisionalization in the esthetic zone: a 1-year randomized controlled prospective study. Int J Oral Maxillofac Implants. 2014 Mar-Apr;29(2):432-40. doi: 10.11607/jomi.3379. PMID 24683571
- [Background] Roe P, Kan JY, Rungcharassaeng K, Caruso JM, Zimmerman G, Mesquida J. Horizontal and vertical dimensional changes of peri-implant facial bone following immediate placement and provisionalization of maxillary anterior single implants: a 1-year cone beam computed tomography study. Int J Oral Maxillofac Implants. 2012 Mar-Apr;27(2):393-400. PMID 22442780
- [Background] van Steenberghe D. Outcomes and their measurement in clinical trials of endosseous oral implants. Ann Periodontol. 1997 Mar;2(1):291-8. doi: 10.1902/annals.1997.2.1.291. PMID 9151562
- [Background] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569
- [Background] Belser UC, Grutter L, Vailati F, Bornstein MM, Weber HP, Buser D. Outcome evaluation of early placed maxillary anterior single-tooth implants using objective esthetic criteria: a cross-sectional, retrospective study in 45 patients with a 2- to 4-year follow-up using pink and white esthetic scores. J Periodontol. 2009 Jan;80(1):140-51. doi: 10.1902/jop.2009.080435. PMID 19228100
- See also: All data can be downloaded from the website, if there are any questions please feel free to contact us. — http://aplicacao.saude.gov.br/plataformabrasil/login.jsf
- Available data/document: Individual Participant Data Set — http://aplicacao.saude.gov.br/plataformabrasil/login.jsf — Public title: Stability of the architecture of the hard and soft tissue after immediate tooth replacement with implants in fresh grafted sockets. All data can be downloaded from the website, if there are any questions please feel free to contact us.
- Available data/document: Study Protocol — http://aplicacao.saude.gov.br/plataformabrasil/login.jsf — Public title: Stability of the architecture of the hard and soft tissue after immediate tooth replacement with implants in fresh grafted sockets. All data can be downloaded from the website, if there are any questions please feel free to contact us.
- Available data/document: Statistical Analysis Plan — http://aplicacao.saude.gov.br/plataformabrasil/login.jsf — Public title: Stability of the architecture of the hard and soft tissue after immediate tooth replacement with implants in fresh grafted sockets. All data can be downloaded from the website, if there are any questions please feel free to contact us.
- Available data/document: Informed Consent Form — http://aplicacao.saude.gov.br/plataformabrasil/login.jsf — Public title: Stability of the architecture of the hard and soft tissue after immediate tooth replacement with implants in fresh grafted sockets. All data can be downloaded from the website, if there are any questions please feel free to contact us.
- Available data/document: Clinical Study Report — http://aplicacao.saude.gov.br/plataformabrasil/login.jsf — Public title: Stability of the architecture of the hard and soft tissue after immediate tooth replacement with implants in fresh grafted sockets. All data can be downloaded from the website, if there are any questions please feel free to contact us.
- Available data/document: Analytic Code — http://aplicacao.saude.gov.br/plataformabrasil/login.jsf — Public title: Stability of the architecture of the hard and soft tissue after immediate tooth replacement with implants in fresh grafted sockets. All data can be downloaded from the website, if there are any questions please feel free to contact us.